CLINICAL TRIAL: NCT05033990
Title: SPIROMICS Study of Early COPD Progression (SOURCE)
Acronym: SOURCE
Status: Recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of North Carolina, Chapel Hill (Other); Columbia University (Other); Johns Hopkins University (Other); National Jewish Health (Other); University of Alabama at Birmingham (Other); University of California, Los Angeles (Other); University of Illinois at Chicago (Other); University of Iowa (Other); University of Michigan (Other); University of Utah (Other); Wake Forest University Health Sciences (Other); Temple University (Other); University of California, San Francisco (Other); COPD Foundation (Other); Weill Medical College of Cornell University (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fernando J Martinez, Professor, University of Massachusetts, Worcester
Other Study IDs: STUDY00002081; R01HL144718 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: COPD, Early-Onset
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, RNA, DNA, exhaled breath condensate, nasal swab, sputum, urine, and stool samples will be collected.
  A subset of participant will undergo bronchoscopy to collect sample such as bronchoalveolar lavage and large and small airway brushings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy Controls: Participants with no smoking history (< 100 cigarettes in lifetime); pre-bronchodilator FEV1/FVC ≥ 0.70; pre-bronchodilator FEV1 ≥ 80% predicted; and pre-bronchodilator FVC ≥ 80% predicted.
- Gold 0: Participants graded as GOLD 0 by the GOLD grading system: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC ≥ 0.70 and FEV1 ≥ 80% predicted.
  GOLD stands for the Global initiative for Chronic Obstructive Lung Disease.
- Preserved Ratio Impaired Spirometry (PRISm): Participants with ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC ≥ 0.70 and FEV1 < 80% predicted.
- GOLD 1 - 2: Participants graded as GOLD 0 by the GOLD grading system: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 ≥ 50% predicted.

SUMMARY:
This is an observational study of 1000 participants to further define the nature of early chronic obstructive pulmonary disease (COPD) in younger, at-risk individuals.

The study has three main goals:

* To use CT scan imaging to identify which smokers will develop COPD.
* To identify biomarkers predictive of smokers that will develop COPD.
* To determine if sputum (phlegm) can be analyzed to predict which smokers will develop COPD.

Procedures (methods): All participants will undergo study related questionnaires assessing medical history, smoke exposure and use, medication use, social and behavioral health, pulmonary symptoms, food frequency, and will provide nasal swab, blood, stool, and urine samples, pulmonary function testing to determine function, sputum induction to provide a sputum sample for airway biospecimen analysis, and CT imaging of the lungs.

ELIGIBILITY:
Inclusion Criteria:

* 40 of the 1000 will be healthy controls: ages 30-55 years; with no smoking history (< 100 cigarettes in lifetime), including vaping and cannabis use; pre-bronchodilator FEV1/FVC > 0.70; pre-bronchodilator FEV1 > 80% predicted; pre-bronchodilator FVC > 80% predicted; Chronic Airway Assessment Test (CAAT) score < 10. Willingness to also participate in the bronchoscopy sub-study is only required of the 20 healthy controls recruited from the clinical centers participating in the sub-study.
* Approximately one-third of the 960 will be GOLD 0 participants: ages 30-55 years; with ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC > 0.70 and FEV1 > 80% predicted.
* Approximately one-third of the 960 will be Preserved Ratio Impaired Spirometry (PRISm) participants: ages 30-55 years; with ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC > 0.70 and FEV1 < 80% predicted.
* Approximately one-third of the 960 will be GOLD 1-2 participants: ages 30-55 years; with ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 > 50% predicted.

Exclusion Criteria:

* Severe asthma, which is defined as any of the following:

  * Current (i.e., at the time of the visit) Global Initiative for Asthma (GINA) Step 4 or higher therapy (medium dose inhaled corticosteroids (ICS)/long-acting beta agonist (LABA) or high dose ICS or add-on long-acting muscarinic agonist (LAMA); Medium dose > 250 fluticasone propionate, = 100 fluticasone furoate, > 200 beclomethasone, > 400 budesonide, > 220 mometasone). We will accept low-dose ICS/LABA or medium dose ICS; or
  * Three or more unscheduled healthcare visits (provider/urgent care/ER) for asthma in the past 12 months; or
  * One asthma hospitalization in the past 12 months.
* Concurrent participation in a therapeutic trial where treatment is blinded.
* Active pregnancy at the time of the baseline visit or planning to become pregnant during the course of the study. This special population is being excluded to minimize potential for fetal radiation exposure.
* Cognitive dysfunction that prevents the participant from completing study procedures.
* BMI > 35.0 kg/m^2 at baseline, due to the effects of body weight on CT scan imaging quality.
* The presence of a respiratory condition other than COPD (including chronic bronchitis and emphysema) or asthma, such as interstitial lung disease or pulmonary fibrosis, or of a comorbid condition that in the judgment of the investigator may be the principal cause of respiratory symptoms (e.g., dyspnea or decreased exercise tolerance).
* Any illness expected to cause mortality in the next three years.
* Any implanted metallic devices or prosthesis above the waist that could degrade thoracic CT scan image quality.
* History of thoracic radiation or thoracic surgery with resection of lung tissue.
* Known HIV/AIDS infection.
* Current illicit substance abuse, excluding marijuana.
* History of or current use of IV Ritalin.
* History of or current use of heroin.
* History of illegal IV drug use within the last 10 years or more than 5 instances of illegal IV drug use ever.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 14 clinical centers across the US will enroll a total of 1000 participants, 30-55 years old, both sexes, all races, and all ethnicities. The participants will include never-smokers (n=40) and GOLD stage 0-2 participants (n=960).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
PRM fSAD | Year 2-5
  Parametric Response Mapping captures the change in lung density between matched inspiratory and expiratory images thereby enabling the distinction between normal lung parenchyma (PRMNORM), emphysema (PRMEMPH), and non-emphysematous air trapping referred to as functional small airway disease (PRMfSAD).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, MS, Principal Investigator — University of Massachusetts Chan Medical School; MeiLan K Han, MD,MS, Principal Investigator — University of Michigan; Jeffrey L Curtis, MD, Principal Investigator — University of Michigan
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Illinois Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Wake Forest, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No